CLINICAL TRIAL: NCT05526053
Title: Preserving Lung Volume During Weaning and Extubation. A Prospective, Multicenter Clinical Trial
Brief Title: Lung Volume Preservation During Extubation
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Althaia Xarxa Assistencial Universitària de Manresa (Other)
Responsible Party: Principal Investigator, Carles Subirà Cuyàs, Research Coordinator, Althaia Xarxa Assistencial Universitària de Manresa
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CEI 22/67
Record Dates: First submitted 2022-08-29; First posted 2022-09-02 (Actual); Last update posted 2025-12-22 (Actual); Status verified 2025-12

CONDITIONS: Weaning Failure; Pulmonary Collapse
Keywords: Weaning from Mechanical Ventilation; Reintubation; Lung Ultrasound Score; Diaphragm and intercostal thickness and thickening fraction
MeSH Terms: conditions — Pulmonary Atelectasis

STUDY DESIGN:
Intervention Model Description: Patients will be allocated to one of the two strategies:
  * Standard OR
  * Preserving Lung volume
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Standard (No Intervention): SBT: PSV 8 cmH2O, PEEP 0 cmH2O for 30 minutes and, when successful, followed by extubation with continuous suctioning.
  Patients included in the ultrasound nested study:
  * Diaphragm and intercostal thickness and thickening fraction at the beginning and the end of the SBT.
  * Modified LUS at the beginning of the SBT, at the end of the SBT and after extubation if successful SBT.
- Lung Volume Preservation (Experimental): SBT: PSV 8 cmH2O, PEEP 5 cmH2O for 30 minutes and, when successful, followed by direct extubation without suctioning and connected to the ventilator with PEEP 5 cmH2O.
  Patients included in the ultrasound part:
  * Diaphragm and intercostal thickness and thickening fraction at the beginning and the end of the SBT.
  * Modified LUS at the beginning of the SBT, at the end of SBT and after extubation if successful SBT.
  Interventions: Other: Lung volume preservation

INTERVENTIONS:
Other: Lung volume preservation — Extubate the patient connected to the ventilator and PEEP of 5 cmH2O after a successful SBT also using PEEP.
  Arms: Lung Volume Preservation

SUMMARY:
Introduction: At present, the best spontaneous breathing trial (SBT) during weaning from mechanical ventilation is a 30-min test with pressure support (PSV) 8 cmH2O without positive end-expiratory pressure (PEEP). There is a debate about the possible collapse of some alveolar units during such SBT and during extubation with continuous suctioning. A few experiences show extubation without suctioning as feasible and safe. Lung ultrasound is a non invasive and useful exploration tool to assess the lung aeration.

Hypothesis: Techniques aimed at preserving lung volume during SBT and extubation can yield higher rates of successful extubation. The preserved lung volume of each SBT and extubation strategy can be assessed by using lung ultrasound.

Primary objective: To define the rates of successful extubation in two extubation approaches aiming at different levels of lung volume preservation: standard SBT (30-min PSV 8 cmH2O without PEEP followed by extubation with continuous suctioning) versus experimental SBT (PSV8+ PEEP 5 cmH2O followed by extubation without suctioning). To define the lung aeration levels using the modified Lung Ultrasound Score (LUS) of each SBT strategy.

Secondary objectives: Reintubation rate, ICU and hospital stays, and mortality in each group. To define the diaphragm and intercostal thickness and thickening fraction in different levels of lung volume preservation.

Design: Prospective, multicenter, randomized study. Two opposing extubation strategies are compared in randomly assigned patients.The level of aeration is assessed using lung ultrasound.

DETAILED DESCRIPTION:
HYPOTHESIS Techniques aimed at preserving lung volume during SBT and extubation can yield higher rates of successful extubation. Lung Ultrasound Score (LUS) might be lower in techniques aiming to preserve lung volume suggesting less lung collapse.

METHODS

Patients with inclusion criteria and none exclusion criteria will be randomized to the follow strategies:

* Standard: PSV 8 cmH2O, PEEP 0 cmH2O for 30 minutes and, when successful, followed by extubation with continuous suctioning.
* Lung volume preservation: PSV 8 cmH2O, PEEP 5 cmH2O for 30 minutes and, when successful, followed by direct extubation without suctioning.

The randomization will be done with the built-in tool of the RedCap® Platform with computerized random number tables and blocks of n patients for each hospital. The investigators of each center will have a profile and a password to log into the RedCap and proceed with randomization of each patient. The investigator of each center will have access only to the data and randomization of his/her center.

In extubation failure patients (those who does not tolerate the SBT or not extubated), the attending physician will decide on the treatment, either support with non-invasive ventilation or with high flow nasal cannula, or reintubation.

Patients who present extubation failure will not be randomized in later SBTs.

During the SBT, interventions that the physician considers necessary to monitor the success of the test, such as echocardiography or thoracic ultrasound, may be performed. In the event that the physician considers that the findings of these tests do not guarantee successful extubation despite fulfillment of extubation criteria according to the study protocol, the attending physician's decision will prevail over the study protocol. In these cases, it will be recorded in the case report form (CRF) as extubation failure due to "other causes of weaning failure".

Not all patients and participating centers will collect data from the lung, diaphragm and intercostal ultrasound assessment. Only those patients that showed interest and proved ultrasound skills, will participate in the ultrasound part of the nested study.

Those patients included in the Ultrasound assessment part, an ultrasonographic exploration will be performed at different times of the SBT and extubation: before starting the SBT, at the final of the SBT and after extubation.

To proof the hypothesis related to the LUS and considering a minimum difference of 1 point (LUSm ranges from 0 to 24 points), we anticipate that 93 in each arm are required .

OBJECTIVES:

Primary: To determine the rate of successful extubation in two opposite weaning strategies.

Secondary:To determine the LUS in two opposite weaning strategies. To determine the ICU stay, hospital stay, hospital survival, and 90-day survival in the two groups. To identify the causes of extubation failure (clinical and ultrasonographic).

Exploratory:To determine the diaphragm and intercostal thickness and thickening fraction in the two groups. To describe patterns of LUS, diaphragmatic and intercostal muscles in patients who fail weaning. To assess changes in LUS during SBT and extubation specifically in posterior-basal regions. To describe diaphragmatic thickening fraction during P0.1 and Pocc maneuvers.

ELIGIBILITY:
Inclusion Criteria:

* Patients> 18 years who meet weaning criteria (see below)
* More than 24 hours of mechanical ventilation (MV)
* Signed Informed Consent by a substitute decision maker (SDM).

Weaning Criteria:

* Suitable cough (Ability to raise secretions to the endotracheal tube) (or Maximal inspiratory pressure (MIP) < -15 cmH2O).
* Absence of excessive secretions (<3 aspirations in the last 8 hours).
* Resolution or improvement of the pathology that led to intubation.
* Clinical stability (Heart Rate (HR) <140 bpm, Systolic Blood Pressure (SBP) 90-160, without vasopressors or at minimum doses).
* Adequate oxygenation (SatO2> 90% with Inspiratory Fraction of oxygen (FiO2) <0.4).
* Adequate ventilatory mechanics (Respiratory rate (RR) <35 rpm, Tidal Volume (TV) > 5 ml / kg, RR / TV <100 rpm/l).
* Confident awareness level (Glasgow Coma Scale (GCS)> 13).

Exclusion Criteria:

* tracheostomy, do-not-reintubate orders, decision of the responsible physician (e.g., due to a preference for a particular weaning technique according to the underlying pathology), absence of informed consent, mental incapacity without legal representation.
* For ultrasound assessment: skilled explorer not present at the time of the SBT, inadequate ultrasound window. Known diaphragmatic paralysis.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1753 (Actual)
Dates: Start 2023-01-15 (Actual); Primary Completion 2024-08-13 (Actual); Study Completion 2024-08-13 (Actual)

PRIMARY OUTCOMES:
Rate of Successful extubation | 72 hours
  Number of patients free of mechanical ventilation

SECONDARY OUTCOMES:
Modified Lung Ultrasound Score (LUSm) at the end of the SBT and after extubation. | 72 hours
  Ultrasound exploration of anterior-superior, anterior-inferior, lateral and posterior-basal. From 0 (no collapse) to 36 (no areation)
Rate of Reintubation | 72 hours
  Number of patients who need reintubation after successful SBT
Rate of ICU Mortality | 90 days
  Patient's Mortality during ICU stay
Rate of Hospital Mortality | 90 days
  Patient's Mortality during hospital stay
Rate of Long term survival | 90 days
  Number of patients alive at 90 days after randomization
ICU length of stay | 90 days
  Mean of days in the ICU
Hospital length of stay | 90 days
  Mean of days in the hospital
Number of patients with tracheostomy | 90 days
  Patients who need tracheostomy
Logistic regression for successful extubation | 90 days
  By using a multilogistic regression, the variables related to successful extubation will be identified.

OTHER OUTCOMES:
Diaphragm thickness at the beginning and at the end of the SBT. | 72 hours
  Maximal thickness measured in M-mode in millimeters.
Diaphragm thickening fraction at the beginning and at the end of the SBT. | 72 hours
  Thickening fraction= (maximal thickness - minimal thickness)/minimal thickness (%)
Intercostal thickness at the beginning and at the end of the SBT. | 72 hours
  Maximal thickness measured in M-mode in millimeters.
Intercostal thickening fraction at the beginning and at the end of the SBT. | 72 hours
  Thickening fraction= (maximal thickness - minimal thickness)/minimal thickness (%)

CONTACTS AND LOCATIONS:
Overall Officials: Rafael Fernandez, PhD, Study Director — Althaia Xarxa Assistencial de Manresa; Carlos Subira, PhD, Principal Investigator — Althaia Xarxa Assitencial de Manresa
Locations (1):
- Althaia Xarxa Assistencial, Manresa, Bacelona, Spain

IPD SHARING:
Plan to Share IPD: No
If any researcher is interested on exploratory analysis, it should be presented to the principal investigator to get the approval for it.

REFERENCES:
- [Background] Brochard L, Rauss A, Benito S, Conti G, Mancebo J, Rekik N, Gasparetto A, Lemaire F. Comparison of three methods of gradual withdrawal from ventilatory support during weaning from mechanical ventilation. Am J Respir Crit Care Med. 1994 Oct;150(4):896-903. doi: 10.1164/ajrccm.150.4.7921460.
- [Background] Esteban A, Alia I, Tobin MJ, Gil A, Gordo F, Vallverdu I, Blanch L, Bonet A, Vazquez A, de Pablo R, Torres A, de La Cal MA, Macias S. Effect of spontaneous breathing trial duration on outcome of attempts to discontinue mechanical ventilation. Spanish Lung Failure Collaborative Group. Am J Respir Crit Care Med. 1999 Feb;159(2):512-8. doi: 10.1164/ajrccm.159.2.9803106. PMID 9927366
- [Background] Esteban A, Alia I, Gordo F, Fernandez R, Solsona JF, Vallverdu I, Macias S, Allegue JM, Blanco J, Carriedo D, Leon M, de la Cal MA, Taboada F, Gonzalez de Velasco J, Palazon E, Carrizosa F, Tomas R, Suarez J, Goldwasser RS. Extubation outcome after spontaneous breathing trials with T-tube or pressure support ventilation. The Spanish Lung Failure Collaborative Group. Am J Respir Crit Care Med. 1997 Aug;156(2 Pt 1):459-65. doi: 10.1164/ajrccm.156.2.9610109. PMID 9279224
- [Background] Perren A, Domenighetti G, Mauri S, Genini F, Vizzardi N. Protocol-directed weaning from mechanical ventilation: clinical outcome in patients randomized for a 30-min or 120-min trial with pressure support ventilation. Intensive Care Med. 2002 Aug;28(8):1058-63. doi: 10.1007/s00134-002-1353-z. Epub 2002 Jul 13. PMID 12185425
- [Background] Esteban A, Anzueto A, Frutos F, Alia I, Brochard L, Stewart TE, Benito S, Epstein SK, Apezteguia C, Nightingale P, Arroliga AC, Tobin MJ; Mechanical Ventilation International Study Group. Characteristics and outcomes in adult patients receiving mechanical ventilation: a 28-day international study. JAMA. 2002 Jan 16;287(3):345-55. doi: 10.1001/jama.287.3.345. PMID 11790214
- [Background] Esteban A, Anzueto A, Alia I, Gordo F, Apezteguia C, Palizas F, Cide D, Goldwaser R, Soto L, Bugedo G, Rodrigo C, Pimentel J, Raimondi G, Tobin MJ. How is mechanical ventilation employed in the intensive care unit? An international utilization review. Am J Respir Crit Care Med. 2000 May;161(5):1450-8. doi: 10.1164/ajrccm.161.5.9902018. PMID 10806138
- [Background] Subira C, Hernandez G, Vazquez A, Rodriguez-Garcia R, Gonzalez-Castro A, Garcia C, Rubio O, Ventura L, Lopez A, de la Torre MC, Keough E, Arauzo V, Hermosa C, Sanchez C, Tizon A, Tenza E, Laborda C, Cabanes S, Lacueva V, Del Mar Fernandez M, Arnau A, Fernandez R. Effect of Pressure Support vs T-Piece Ventilation Strategies During Spontaneous Breathing Trials on Successful Extubation Among Patients Receiving Mechanical Ventilation: A Randomized Clinical Trial. JAMA. 2019 Jun 11;321(22):2175-2182. doi: 10.1001/jama.2019.7234. PMID 31184740
- [Background] Fernandez MM, Gonzalez-Castro A, Magret M, Bouza MT, Ibanez M, Garcia C, Balerdi B, Mas A, Arauzo V, Anon JM, Ruiz F, Ferreres J, Tomas R, Alabert M, Tizon AI, Altaba S, Llamas N, Fernandez R. Reconnection to mechanical ventilation for 1 h after a successful spontaneous breathing trial reduces reintubation in critically ill patients: a multicenter randomized controlled trial. Intensive Care Med. 2017 Nov;43(11):1660-1667. doi: 10.1007/s00134-017-4911-0. Epub 2017 Sep 22. PMID 28936675
- [Result] Andreu M, Bertozzi M, Bezzi M, Borello S, Castro D, Giorgio VD, Aguirre M; ExtubAR group; ExtubAR group is composed by. Comparison of Two Extubation Techniques in Critically Ill Adult Subjects: The ExtubAR Randomized Clinical Trial. Respir Care. 2022 Jan;67(1):76-86. doi: 10.4187/respcare.09276. Epub 2021 Nov 3. PMID 34732586
- [Result] Soummer A, Perbet S, Brisson H, Arbelot C, Constantin JM, Lu Q, Rouby JJ; Lung Ultrasound Study Group. Ultrasound assessment of lung aeration loss during a successful weaning trial predicts postextubation distress*. Crit Care Med. 2012 Jul;40(7):2064-72. doi: 10.1097/CCM.0b013e31824e68ae. PMID 22584759
- [Result] Tenza-Lozano E, Llamas-Alvarez A, Jaimez-Navarro E, Fernandez-Sanchez J. Lung and diaphragm ultrasound as predictors of success in weaning from mechanical ventilation. Crit Ultrasound J. 2018 Jun 18;10(1):12. doi: 10.1186/s13089-018-0094-3. PMID 29911284
- [Derived] Subira C, Rognoni G, Baquerizo H, Garcia C, Cabanes S, de la Torre M, Quevedo B, Pedros C, Tizon AI, Murillo N, Parro L, Eiras F, Rialp G, Altaba S, Gonzalez-Castro A, Pacheco AF, Bayoumi P, Gomez-Medrano N, Vallverdu I, Higon A, Navarro MD, Falcon A, Keough E, Arizo D, Martinez JF, Duran N, Rodriguez R, Popoviciu-Koborzan MR, Guerrero I, Concha P, Barral P, Batlle M, Cano S, Garcia-Castrillon S, Andorra X, Tua Y, Arnau A, Fernandez R. Effect of lung volume preservation during spontaneous breathing trial on successful extubation in patients receiving mechanical ventilation: protocol for a multicenter clinical trial. Trials. 2024 Jul 16;25(1):481. doi: 10.1186/s13063-024-08297-1. PMID 39014430

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2023-04-26): https://cdn.clinicaltrials.gov/large-docs/53/NCT05526053/Prot_SAP_002.pdf
  • Informed Consent Form (2022-08-26): https://cdn.clinicaltrials.gov/large-docs/53/NCT05526053/ICF_001.pdf